CLINICAL TRIAL: NCT01561118
Title: DiaSport - Ausdauerorientiertes Trainingsprogramm Mit Kindern Und Jugendlichen an Der Dialyse (DiaSport - Endurance-orientated Training Program With Children and Adolescents on Maintenance Hemodialysis)
Brief Title: DiaSport - Endurance-orientated Training Program With Children and Adolescents on Maintenance Hemodialysis
Acronym: DiaSport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. B. Hoppe, Prof. Dr. med., University of Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Uni-Koeln-1137; DFG HO 1272/21-1 (Other Grant/Funding Number: DFG HO 1272/21-1)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: hemodialysis; dialysis efficacy; cardiorespiratory capacity; exercise capacity; children and adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicycle-Ergometer Training Group (Experimental): Performance adapted, hence individualised three times weekly bicycle-ergometer training during hemodialysis. Each training will last 30 to 50 minutes, with 70-80% of the patient specific maximum workload over 12 weeks (36 training sessions).
  In the second part of the study intervention will be prolonged for another 12 weeks.
  Interventions: Other: Bicycle-Ergometer Training
- Control (Other): No intervention during hemodialysis during the first 12 weeks of the study.
  In the second part of the study a training program, according to that of the intervention group, will be performed with a performance adapted, hence individualised three times weekly bicycle-ergometer training during hemodialysis. Each training will last 30 to 50 minutes, with 70-80% of the patient specific maximum workload over 12 weeks (36 training sessions).
  Interventions: Other: Bicycle-Ergometer Training

INTERVENTIONS:
Other: Bicycle-Ergometer Training — Performance adapted, hence individualised three times weekly bicycle-ergometer training during hemodialysis. Each training will last 30 to 50 minutes with 70-80% of the patient specific maximum workload over 12 weeks (36 training sessions - first part of the study compared to no intervention).
  In the second part of the study both groups get the opportunity for another 12 weeks of individualised three times weekly bicycle-ergometer training during hemodialysis.

SUMMARY:
Physical activity is considered essential for optimal health, development, socialization and well-being of children. However patients with end-stage renal disease (ESRD) are often restricted from participation in exercise activities. This is especially true for children on hemodialysis (HD). As a consequence their exercise capacity is reduced, both before, but most impressively after HD. In a nationwide randomized, multi-center design this study aims to proof the influence of an individualised endurance training program by bicycle ergometer performed during dialysis on the efficacy of HD, measured as single pool Kt/V. Secondary goals are to enhance physical performance, physical and mental well-being, and to improve measurable blood and treatment parameters (e.g. haemoglobin level, amount of medication). A positive impact of physical activity was observed in adults on HD, although most studies did not address this issue in a randomised protocol. Despite this beneficial evidence in adults, sport is still not integrated as part of standard care in patients on maintenance HD. The study protocol, developed in close collaboration with the German Sport University Cologne, differs substantially from previously published reports as it uses bicycle ergometer training in an upright position outside the dialysis couch and adapts the intensity of intervention to the patient's capabilities. Based on the expected results the investigators will develop an individualised training program to be integrated in the standard care of (pediatric) patients on maintenance HD.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease with need of renal replacement therapy
* children and adolescents aged ≥6 to ≤19 years
* maintenance hemodialysis for at least 3 months
* Stable and appropriate dialysis condition in the last 4 weeks before inclusion to the study (basically stable blood and dialysate flow rate and same dialyser)
* single pool Kt/V according to Dialysestandard 2006 > 1.2
* Informed consent

Exclusion Criteria:

* Participation in another interventional clinical trial
* severe primary neurologic, orthopaedic or cardiac disease, or secondary disease known as a contraindication for endurance training
* uncontrolled hyper- or hypotension, or cardiac disease
* Recurrent uncontrolled epileptic seizures
* dialysis shunt at the lower limbs
* pregnancy
* already planned medical intervention, for example living donor kidney transplantation or any other surgery, within the first period of the trial which will cause cancelation of more then 3 training units in a row
* Subjects who are in dependency to the sponsor or the PI of the trial, or confined to an institution on judicial or official behalf

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change of single pool Kt/V (KDOQI Guidelines) - expressed as the change of single pool Kt/V from week 0 to 12 of intervention (period 1) | 12 weeks
  Change of single pool Kt/V (spKt/V) measured at week 12 (V1) compared to baseline (V0). Single pool Kt/V is the standard measure to assess dialysis efficacy. As dialysis efficacy is the primary aim of dialysis treatment and the spKt/V is the best way to measure efficacy this figure has an important clinical relevance for the patient.

SECONDARY OUTCOMES:
Change of the possible workload (maximum physical performance) achieved | 12 and 24 weeks
  The maximal possible workload will be determined by an exercise evaluation program with increasing power on a leg bicycle ergometer before a hemodialysis session, measuring the peak oxygen uptake (VO2-peak), heart rate, blood pressure and lactate levels during exercise.
Quality of Life | 12 and 24 weeks
  For quality of life assessment the validated and standardized PedsQL® questionnaires will be filled in by patients and parents.
Change of solute removal during hemodialysis | 12 and 24 weeks
  Solute removal during hemodialysis has a clear impact on the patient's health and well-being, as it reduces sequelae and offers the patient less restrictions on their diet, which would lead to a better compliance.
Change of solute removal in the two compartment model (assessed in a subgroup of patients) | 12 and 24 weeks
  Solute removal in the two compartment model will only be analyzed in patients 12 years of age or older with explicit consent to a second blood drawing 30 minutes after end of hemodialysis session. It was previously used showing a significant enhancement during exercise, explained by an increase of skeletal muscles perfusion during exercise.
Inflammation, nutritional status and bone metabolism | 12 and 24 weeks
  The nutritional status and bone metabolism will be determined as they are important for optimal health and growth of paediatric hemodialysis patients. Evidence is based on studies that showed trends towards a better nutritional status and less chronic inflammation.
Body Composition Monitoring (BCM) | 12 and 24 weeks
  Body Cpomposition Monitoring (BCM) will be performed to exermine further information on nutrional status, overhydration and muscle growth.
Change of number and dose of medication needed | 12 and 24 weeks
  Number and dose of medication will be recorded, changes will be evaluated, and data will be correlated to e.g. the measured blood pressure (antihypertensive drugs) or haemoglobin levels (EPO or EPO stimulating agents).
Telomere length and Telomerase activity | 12 and 24 weeks
  Telomere length and telomerase activity [units] will be used as markers for cell survival, which may be influenced by endurance training.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hoppe, MD, Study Chair — University Hospital of Bonn; Bettina Schaar, PhD, Study Chair — German Sport University, Cologne
Locations (1):
- University Hospital Bonn. Department of Pediatric and Adolescent Medicine, Division of Pediatric Nephrology, Bonn, Germany

REFERENCES:
- [Background] Schaar B, Feldkotter M, Nonn JM, Hoppe B. Cardiorespiratory capacity in children and adolescents on maintenance haemodialysis. Nephrol Dial Transplant. 2011 Nov;26(11):3701-8. doi: 10.1093/ndt/gfr014. Epub 2011 Mar 4. PMID 21378148
- [Background] Hoppe B, Schaar B. The impact of nutrition and physical activity on long-term survival after pediatric solid organ transplantation. Pediatr Transplant. 2012 Nov;16(7):675-7. doi: 10.1111/j.1399-3046.2012.01663.x. Epub 2012 Feb 21. No abstract available. PMID 22353206
- [Derived] Feldkotter M, Thys S, Adams A, Becker I, Buscher R, Pohl M, Schild R, Pape L, Schmitt CP, Taylan C, Wygoda S, Klaus G, Fehrenbach H, Montoya C, Konrad M, Billing H, Schaar B, Hoppe B. Endurance-oriented training program with children and adolescents on maintenance hemodialysis to enhance dialysis efficacy-DiaSport. Pediatr Nephrol. 2021 Dec;36(12):3923-3932. doi: 10.1007/s00467-021-05114-8. Epub 2021 Jun 12. PMID 34117528